CLINICAL TRIAL: NCT06401044
Title: A Phase 1/2, Randomized, Double-Masked, Placebo-Controlled, Multicenter Study to Assess the Safety, Pharmacokinetics, and Efficacy of AMG 732 in Healthy Subjects and Subjects With Moderate-to-Severe Active Thyroid Eye Disease
Brief Title: A Study of AMG 732 in Healthy Participants and Participants With Thyroid Eye Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20230302
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease
Keywords: AMG 732; Thyroid Eye Disease; TED
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: AMG 732 (Experimental): Participants in 6 cohorts will receive either AMG 732 or placebo in Single Ascending Doses (SAD).
  Interventions: Drug: AMG 732
- Part A: Placebo (Placebo Comparator): Participants in 6 cohorts will receive either AMG 732 or placebo in Single Ascending Doses (SAD).
  Interventions: Other: Placebo
- Part B: AMG 732 Low Dose (Experimental): Participants will receive AMG 732 low dose SC.
  Interventions: Drug: AMG 732
- Part B: AMG 732 Medium Dose (Experimental): Participants will receive AMG 732 medium dose SC.
  Interventions: Drug: AMG 732
- Part B: AMG 732 High Dose (Experimental): Participants will receive AMG 732 high dose SC.
  Interventions: Drug: AMG 732
- Part B: Placebo (Placebo Comparator): Participants will receive placebo SC.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AMG 732 — SC injection
  Arms: Part A: AMG 732; Part B: AMG 732 High Dose; Part B: AMG 732 Low Dose; Part B: AMG 732 Medium Dose
Other: Placebo — SC injection
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The primary objective of Part A of this study is to investigate the safety and tolerability of AMG 732 after single subcutaneous (SC) doses. The primary objective of Part B of this study is to investigate the efficacy of AMG 732 in participants with Thyroid Eye Disease (TED) after multiple SC doses.

DETAILED DESCRIPTION:
Recruitment has ended for the Phase 1 portion of the study and will reopen when Phase 2 begins recruitment.

ELIGIBILITY:
Inclusion criteria for Part A/Phase 1 only:

* Participant has provided informed consent before initiation of any study-specific activities/procedures.
* Male or female aged 18 to 55 years (Part A).
* Female participants must be of non-childbearing potential.
* Body mass index (BMI) between 18 and 30 kg/m^2, inclusive, at screening.
* The participant has adequate venous access and can receive intravenous (IV) therapy.
* The participant is considered by the investigator or designee to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at screening.
* Healthy Japanese participants in cohort 4 only. Japanese participants must meet all the following as confirmed by interview: Descendants of 4 ethnic Japanese grandparents who were born in Japan; Both parents are ethnic Japanese who were born in Japan; Hold a Japanese passport or identity papers; Have lived outside Japan for less than 10 years at the time of screening and lifestyle including diet has not changed significantly since leaving Japan.

Inclusion criteria for Part B/Phase 2 only:

* Male or female aged 18 to 65 years.
* Moderate-to-severe active TED.
* The participant had onset of active TED within 15 months prior to baseline.
* Clinical diagnosis of Graves' disease associated with active TED with a Clinical Activity Score (CAS)≥3 for the most severely affected eye at screening and baseline.
* Proptosis ≥18mm in the study eye at baseline.
* Participants with baseline subjective binocular diplopia score >0.
* Does not require immediate surgical ophthalmological intervention and is not planning corrective surgery/irradiation during the trial.

Exclusion criteria for Part A and Part B:

* Malignant condition in the past 12 months or major surgery within 8 weeks or plans to have an elective surgery from screening through end of study.
* Active liver or kidney disfunction at screening.
* Positive test for hepatitis B/C or Human immunodeficiency virus (HIV) serology at screening.
* Glycated hemoglobin (HbA1c) > 6.5% and/or fasting glucose levels> 126 mg/dL (> 7 mmol/L) at screening.
* Use of any steroid (IV, oral, steroid eye drops) within 3 weeks prior to the first dose. Steroids cannot be initiated during the trial. Exceptions include topical and inhaled steroids and steroids used to treat injection related reactions or short course of steroid for asthma control.
* Known hypersensitivity to teprotumumab or any other monoclonal antibody products.
* History of substance abuse within 12 months before screening.
* Donated blood, or had significant blood loss, or received a transfusion of any blood or blood products within 60 days prior to day 1 dosing or received a plasma donation within 7 days prior to day 1 dosing.

Exclusion criteria for PartA/Phase 1 only

• Blood pressure or ECG abnormalities at screening.

Exclusion criteria for Part B/Phase 2 only:

* Use of any steroid or other non-steroid immunosuppressive agent, monoclonal antibody, within 3 months prior to the first injection of study drug.
* Use of teprotumumab or any other IGF-1R inhibitor.
* Prior orbital irradiation or decompression in the study eye.
* History or existing inflammatory bowel disease (ulcerative colitis or Crohn's disease).

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-08-13 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of Participants With Treatment-emergent Adverse Events | Day 1 through Week 36 (End of Study)
Part B: Change from Baseline in Proptosis Measurement by an Exophthalmometer in the Study Eye | Baseline to End of Treatment (EoT) (approximately 6 Months)

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of AMG 732 | Up to Week 36
Part A: Time to Cmax (Tmax) of AMG 732 | Up to Week 36
Part A: Area Under the Plasma Concentration-time Curve (AUC) of AMG 732 | Up to Week 36
Part A: Half-life (t1/2) of AMG 732 | Up to Week 36
Part A: Number of Participants With Anti-drug Antibodies (ADAs) | Up to Week 36
Part B: Number of Participants With Treatment-emergent Adverse Events | Up to Week 48
Part B: Cmax of AMG 732 | Up to Week 48
Part B: Tmax of AMG 732 | Up to Week 48
Part B: AUC of AMG 732 Over the Dosing Interval | Up to Week 48
Part B: Accumulation of AMG 732 Following Multiple Dosing | Up to Week 48
Part B: Half-life (t1/2) of AMG 732 | Up to Week 48
Part B: Number of Participants With Anti-drug Antibodies (ADAs) | Up to Week 48
Part B: Proptosis Response Status in the Study Eye | EoT (approximately 6 Months)
Part B: Mean Change from Baseline in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Visual Functioning (VF) Subscale Score | Baseline to EoT (approximately 6 Months)
Part B: Mean Change from Baseline in the GO-QoL Appearance (A) Subscale Score | Baseline to EoT (approximately 6 Months)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- United States (9):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Levenson Eye Associates, Jacksonville, Florida
  - Ilumina Medical Research, Kissimmee, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Vision Medical Research, Inc., Orland Park, Illinois
  - Ppd Las Vegas Research Unit, Las Vegas, Nevada
  - Erie Retina Research, Erie, Pennsylvania
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - West Virginia University, Morgantown, West Virginia
- Australia (2):
  - Macquarie University, North Ryde, New South Wales
  - North Shore Private Hospital, St Leonards, New South Wales
- Vancouver General Hospital, Vancouver, British Columbia, Canada
- France (2):
  - Centre Hospitalier Universitaire de Nantes - Hopital Nord Laennec, Nantes
  - Hopital Pitie-Salpetriere, Paris
- Universitaetsklinikum Essen, Essen, Germany
- Poland (2):
  - Dc-Med Spolka z Ograniczona Odpowiedzialnoscia Spolka Komandytowa, Swidnica
  - Eb Group Spolka z ograniczona odpowiedzialnoscia, Warsaw
- Singapore National Eye Centre, Singapore, Singapore
- Spain (3):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com